CLINICAL TRIAL: NCT04713280
Title: Maxillary Versus Bi-Maxillary Posterior Segments Intrusion in Treatment of Adult Subjects With Skeletal Open Bite - A Randomized Clinical Trial
Brief Title: Maxillary Versus Bi-Maxillary Posterior Segments Intrusion Adult Subjects With Skeletal Open Bite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba El-Sayed Kamel Akl, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2098765
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Dental Malocclusion
Keywords: molar intrusion; open bite; mini-screws
MeSH Terms: conditions — Malocclusion; Open Bite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxillary posterior dento-alveolar intrusion (Active Comparator): Mini-screw supported maxillary posterior dento-alveolar intrusion
  Interventions: Procedure: Maxillary posterior dento-alveolar intrusion
- Bi-maxillary posterior dento-alveolar intrusion (Experimental): Mini-screw supported bi-maxillary posterior dento-alveolar intrusion
  Interventions: Procedure: Maxillary posterior dento-alveolar intrusion

INTERVENTIONS:
Procedure: Maxillary posterior dento-alveolar intrusion — Mini-screw supported maxillary or bi-maxillary posterior dento-alveolar intrusion
  Other Names: Bi-maxillary posterior dento-alveolar intrusion

SUMMARY:
Compare between bi-maxillary (maxillary and mandibular) posterior dento-alveolar intrusion and maxillary posterior dento-alveolar intrusion as regards open bite closure.

DETAILED DESCRIPTION:
Now, maxillary posterior dento-alveolar intrusion has been validated as a conservative treatment modality for treatment of skeletal open bite in adult patients. However, it was proved that mandibular posterior teeth extrusion take place during the treatment which results in reduction in the amount of open. bite closure. Therefore, the aim of our study is to compare in a randomized clinical trial methodology between maxillary posterior dento-alveolar intrusion and combined maxillary and mandibular posterior dento-alveolar intrusion in terms of anterior open bite closure.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal open bite with a dental open bite ranging from 3-8 mm.
* Adequate incisal show at rest and on smiling
* Full set of posterior teeth from first premolar to second molar (with the exception of one tooth in one quadrant).

Exclusion Criteria:

* Dental open bites without skeletal components
* Previous orthodontic treatment
* Medically compromised patients

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Anterior open bite closure | 6 months
  The amount of overbite gained as a result of posterior dento-alveolar intrusion

SECONDARY OUTCOMES:
Maxillary posterior teeth intrusion radiographically in millimeters. | 6 months
  The distance travelled by maxillary premolars and molars of the right and left sides to a reference plane
Mandibular posterior teeth intrusion radiographically in millimeters. | 6 months
  The distance travelled by mandibular premolars and molars of the right and left sides to a reference plane
Tip and torque of intruded teeth radiographically in degrees. | 6 months
  • Torque change is measured as the change in the angle between the long axis of the intruded teeth and the FH plane (for tip) mid-sagittal plane (for torque).

CONTACTS AND LOCATIONS:
Overall Officials: Heba Akl, MSc., Principal Investigator — Assistant lecturer, PhD candidate
Locations (1):
- Orthodontic Department, Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Akl HE, Abouelezz AM, El Sharaby FA, Abd-El-Ghafour M, El-Beialy AR. Is mandibular posterior dento-alveolar intrusion essential in treatment of skeletal open bite in adult patients? A single center randomized clinical trial. BMC Oral Health. 2025 Apr 7;25(1):500. doi: 10.1186/s12903-025-05778-w. PMID 40197278